CLINICAL TRIAL: NCT05968014
Title: Quality of Recovery After Hip Fracture Surgery: Ultrasound-guided Pericapsular Nerve Group Block Versus Fascia Iliaca Compartment Block
Brief Title: Quality of Recovery After Hip Fracture Surgery: US-guided PENG Block Versus FICB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Chaima Debabi, Principal Investigator, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Chaima Debabi
Record Dates: First submitted 2023-07-11; First posted 2023-08-01 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2023-07

CONDITIONS: Enhanced Recovery After Surgery
Keywords: hip fracture surgery; PENG block; fascia iliaca compartment block; quality of recovery

STUDY DESIGN:
Intervention Model Description: randomised-controlled trial with two parallel study groups. Participants will be randomised 1:1 to the PENG group or FICB group. The PENG group was treated with PENG block following randomisation, whereas the FICB group received a fascia iliaca compartment block.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG block (Experimental): Participants enrolled in this group received a pericapsular nerve group block with 20 ml of 0.2% ropivacaine. The block was performed with a 100 mm needle, inserted with an in-plane lateral to medial approach. Operator used a low frequency curvilinear probe.
  Interventions: Procedure: PENG vs FICB
- FIC block (Experimental): Patients allocated in this group received a fascia iliaca compartment block with 20 mL of 0.2% ropivacaine, using a 50 mm needle inserted with an in-plane approach. Operator used a linear probe.
  Interventions: Procedure: PENG vs FICB

INTERVENTIONS:
Procedure: PENG vs FICB — pericapsular nerve group block versus fascia iliaca compartment block

SUMMARY:
Patients were randomly divided into two groups to receive either ultrasound-guided pericapsular nerve group block (PENG group) or fascia iliaca compartment block (FICB group), using 20 ml of 0.2% ropivacaine

DETAILED DESCRIPTION:
Participants were randomly divided into two groups : group PENG and group FICB, to receive either ultrasound-guided pericapsular nerve group block or fascia iliaca compartment block, using 50 ml of 0.2% ropivacaine.

For the FICB, a linear ultrasound probe was placed in the transverse plane and start scanning at the level of the inguinal crease to identify the femoral artery medially and the femoral nerve lateral to the femoral artery. The iliopsoas muscle should be seen overlying fascia iliaca. The block should be performed proximal to the arterial bifurcation. A 50 mm needle was introduced using an in-plane approach to penetrate the fascia iliaca. The hydro dissection separate the fascia iliaca from the iliac muscle, and a total volume of 20 ml of 0.2% ropivacaine was injected in this created space.

The PENG bloc is performed with a low frequency curvilinear ultrasound probe, which was initially placed in a transverse plane over the antero inferior iliac spine and the aligned with the pubic ramus by rotating the probe counterclockwise approximately 45 degrees. In this view, it is possible to observe the iliopubic eminence, the iliopsoas muscle tendon, the femoral artery and the pectineus muscle. A 100 mm needle was inserted from lateral to medial in an in-plane approach to place the tip in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly. Negative aspiration should be observed before injection of local anaesthetic and a total volume of 20 ml of 0.2% ropivacaine was injected.

Spinal anesthesia was performed after 20 minutes.

QoR-15 score was assessed before the intervention and 24 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* patients aged above 65 years
* patients with an american society of anesthesiologists physical status I to III
* patients undergoing hip fracture surgical repair

Exclusion Criteria:

* patients with an american society of anesthesiologists physical status IV or more
* inability or refusal to sign informed consent
* contraindications for regional nerve block or spinal anesthesia
* impaired cognition or dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
The Quality of Recovery-15 scores at 24 hours postoperatively. | before and 24 hours after surgery
  Change in Quality of Recovery-15 (QoR-15) scores before and 24 hours after surgery.
  The QoR-15 score consists of 15 items, and includes five dimensions: pain (two items), physical confort (five items), physical independance (two items), psychological support (two items) and emotional state (four items). Each item's score ranged from 0 to 10, and the total score ranged from 0 to 150, with a higher QoR-15 score indicating a better quality of recovery.

SECONDARY OUTCOMES:
The strength of the quadriceps | 24 hours after surgery
  The strength of the quadriceps muscle was measured 24 hours after surgery. It was determined by testing the movement of the knee and the hip.
Visual analogue scale | 24 hours after surgery
  change in visual analogue scale ((VAS) with 0 indicating no pain and 10 indicating the worst imaginable pain) at rest and on movement on postoperative day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Chaima Debabi, Principal Investigator — University Tunis El Manar
Locations (1):
- Nabeul hospital, Mohamed Taher Maamouri, Nabeul, Mrezga, Tunisia

IPD SHARING:
Plan to Share IPD: No